CLINICAL TRIAL: NCT03839433
Title: Ciclesonide for the Treatment of Airway Hyperresponsiveness: The Mannitol-Asthma-Ciclesonide-Study
Brief Title: The Mannitol-Asthma-Ciclesonide-Study
Acronym: MACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Prof. Dr., Cantonal Hosptal, Baselland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY 9010 / CH-101
Record Dates: First submitted 2017-08-04; First posted 2019-02-15 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Asthma, Bronchial
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ciclesonide positive (Active Comparator): Half of the Mannitol positive patients were given ciclesonide. Half of the Mannitol negative patients were given ciclesonide. All patients in the "ciclesonide positive" arm received ciclesonide.
  Interventions: Drug: Ciclesonide
- Placebo (Placebo Comparator): Half of the Mannitol positive patients were given a placebo. Half of the Mannitol negative patients were given a placebo. All patients in the "placebo" arm received placebo.
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
Response of a 4 weeks treatment with daily once 320 µg ciclesonide on airway hyperresponsiveness assessed with mannitol.

Hypothesis: Treatment with inhaled ciclesonide reduces airway hyper-responsiveness in 80% of hyper-responsive patients compared to 20% only in the placebo group and the group without airway hyper-responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the pulmonology department of the university hospital Basel because of suspected asthma defined as respiratory symptoms like wheezing or cough or chest tightness.
* Asthma symptoms partly controlled according to GINA (Global Initiative for Asthma, October 2006) 1 week prior to randomization
* FEV1 ≥ 70% predicted

Exclusion Criteria:

* Smoker and ex-smoker with >10 pack years
* COPD (chronic obstructive pulmonary disease)
* Upper respiratory tract infection within the past 4 weeks.
* ICS or oral steroids during the previous month before inclusion
* beta-blockers within the past 4 weeks
* Current treatment with medication as defined in section concomitant medication (ICS other than study medication, ß-blockers)
* Pregnancy
* Known malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change of hyperresponsiveness to mannitol by measuring PD15 FEV1 after 4 weeks (improvement of more than at least 1.5 doubling dose) | 4 weeks
  measurements of PD15 FEV1 (provocative dose to produce a 15% fall in FEV1), bronchial hyperresponsiveness. A 15 % reduction of FEV1 means a bronchial hyperresponsiveness

SECONDARY OUTCOMES:
Change in PD20 FEV1 methacholine (Responsiveness to metacholine) | 4 weeks
  measurements of PD20 FEV1 (provocative dose to produce a 20% fall in FEV1) bronchial hyperresponsiveness. A 20 % reduction of FEV1 means a bronchial hyperresponsiveness
Change in FeNO (Nitric Oxide) | 4 weeks
  Measurement of bronchial inflammation. It determines the level of nitric oxide in parts per billion (PPB). Nitric oxide in exhaled air is another marker of airway inflammation. Subjects with atopic asthma or rhinitis seem to have elevated expiratory nitric oxide (eNO) levels.
Change in ACQ (Asthma Control Questionnaire) | 4 weeks
  It measures both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment. It measures both the adequacy of asthma control and change in asthma control, which occurs either spontaneously or as a result of treatment. The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% pred. and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
AQLQ (Asthma Quality of Life Questionnaire) | 4 weeks
  The Asthma Quality of Life Questionnaire (AQLQ) was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults (17-70 years) with asthma. There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). The activity domain contains 5 'patient-specific' questions. This allows patients to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.